CLINICAL TRIAL: NCT04278885
Title: Factor XII-associated Cold Autoinflammatory Syndrome (FACAS) Linked to Kallikrein-kinin Pathology: Proof of Concept Treatment With Lanadelumab (DX-2930)
Brief Title: Lanadelumab in FXII-associated Cold Autoinflammatory Syndrome (FACAS)
Acronym: LANA-FXII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Shire International GmbH (Unknown)
Responsible Party: Principal Investigator, Karoline Krause, Professor, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEALSZ-2019-01
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Hereditary Autoinflammatory Disease
Keywords: FXII-associated cold autoinflammatory syndrome (FACAS)
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases | interventions — lanadelumab

STUDY DESIGN:
Intervention Model Description: exploratory, proof-of-concept, single-center, open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lanadelumab (Experimental)
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — 300mg Lanadelumab s.c. administration every 2 weeks
  Other Names: DX-2930

SUMMARY:
This is a Phase 2, exploratory, proof-of-concept, single-center, open-label pilot study to assess the effects and safety of Lanadelumab in patients with FXII-associated cold autoinflammatory syndrome (FACAS).

DETAILED DESCRIPTION:
Factor XII is a serine protease with diverse functions that participates in coagulation, fibrinolysis, complement and contact system activation. So far, mutations in the factor XII gene were linked to the rare coagulation disorder Hagemann factor deficiency and hereditary angioedema (FXII-HAE).

The investigators recently identified a novel FXII mutation in a 4-generation family with profound contact system activation and an autoinflammatory clinical phenotype.

Lanadelumab is a specific kallikrein Inhibitor that is known to prevent clinical symptoms and contact system activation in hereditary angioedema.

This study aims at assessing the clinical effects and safety of Lanadelumab in patients with FXII-associated cold autoinflammatory syndrome (FACAS).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (12 - 17 years) and adults (18 years or older)
* Documented FXII-associated autoinflammatory disorder (FACAS) by positive genetic analysis result
* Clinical symptoms of cold-associated wheals, arthralgia, headache, fatigue (FACAS)
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* Males and females who are fertile and sexually active must adhere to contraception requirements for the duration of the study as follows:
* Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception from the screening period through 30 days after the final study visit: progestin-only oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD, all types). Female participants whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
* Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
* Males, including males who are surgically sterile (post vasectomy), with female partners of childbearing potential must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the last IMP injection.

Exclusion Criteria:

* 1. Any other forms of urticaria or angioedema not related to genetic mutations within the FXII gene 2. Concurrent/ongoing treatment with biologics or recent treatment (less than 5 half-lives) 3. Concurrent/ongoing treatment with anakinra within 7 days prior to screening, with canakinumab within 100 days prior to screening 4. Concurrent/ongoing treatment with oral/parenteral corticosteroids greater than 10 mg/d within 2 weeks prior to screening 5. Concurrent/ongoing treatment with other immunosuppressives within 4 weeks or 5 half-lives prior to screening, whichever is longer 6. Treatment with a live (attenuated) virus vaccine within 4 weeks prior to Baseline visit 7. Exposure to angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications with systemic absorption (such as oral contraceptives or hormonal replacement therapy) within 4 weeks prior to screening.

  8. Use of prophylactic therapy with C1-INH, attenuated androgens, or antifibrinolytics within 2 weeks prior to the start of the treatment period (Day 0).

  9. Any of the following liver function test abnormalities:
  * alanine aminotransferase (ALT) > 3x upper limit of normal, or
  * aspartate aminotransferase (AST) > 3x upper limit of normal, or
  * total bilirubin > 2x upper limit of normal (unless the bilirubin elevation is a result of Gilbert's Syndrome).

    10. Pregnancy or breastfeeding. 11. Subject has any condition that, in the opinion of the Investigator or Sponsor, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (e.g., history of substance abuse or dependence, a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of study results).

    12. Significant medical condition rendering the patient immunocompromised or not suitable for a clinical trial.

    13. Enrollment in another investigational treatment or device study or use of an investigational agent, or less than 4 weeks or 5 half-lives, whichever is longer, since end of another investigational device or drug trial.

    14. Patients with known hypersensitivity to any constituent of the products of lanadelumab.

    15. Dementia, altered mental status, or any psychiatric condition, or stay in an institution further to an official or court order that would prohibit the understanding or rendering of informed consent or participation in the study.

    16. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in total disease activity score as assessed by daily health assessment form (DHAF) questionnaire following lanadelumab treatment | weeks 9 to 12 compared to weeks -4 to -1 (baseline)
  Patient-reported total disease activity is assessed by a disease-specific daily health assessment form (FXII-associated Cold autoinflammatory Syndrome daily Health assessment form; FACAS-DHAF) grading the severity of 5 key symptoms of FACAS: urticarial rash, fatigue, chills/fever, arthralgia and headache (scale 0=no symptoms to 50=max. of symptoms).

SECONDARY OUTCOMES:
Change in urticarial rash disease activity score as assessed by daily health assessment form (DHAF) questionnaire following lanadelumab treatment | weeks 9 to 12 and weeks 24 to 28, each compared to weeks -4 to -1 (baseline)
  Patient-reported urticarial rash disease activity is assessed by a disease-specific daily health assessment form (FXII-associated Cold autoinflammatory Syndrome daily Health assessment form; FACAS-DHAF; scale 0=no symptoms to 10=max. of symptoms)
Change in fatigue disease activity score as assessed by daily health assessment form (DHAF) questionnaire following lanadelumab treatment | weeks 9 to 12 and weeks 24 to 28, each compared to weeks -4 to -1 (baseline)
  Patient-reported fatigue disease activity is assessed by a disease-specific daily health assessment form (FXII-associated Cold autoinflammatory Syndrome daily Health assessment form; FACAS-DHAF; scale 0=no symptoms to 10=max. of symptoms)
Change in chills/fever disease activity score as assessed by daily health assessment form (DHAF) questionnaire following lanadelumab treatment | weeks 9 to 12 and weeks 24 to 28, each compared to weeks -4 to -1 (baseline)
  Patient-reported chills/fever disease activity is assessed by a disease-specific daily health assessment form (FXII-associated Cold autoinflammatory Syndrome daily Health assessment form; FACAS-DHAF;scale 0=no symptoms to 10=max. of symptoms)
Change in arthralgia disease activity score as assessed by daily health assessment form (DHAF) questionnaire following lanadelumab treatment | weeks 9 to 12 and weeks 24 to 28, each compared to weeks -4 to -1 (baseline)
  Patient-reported arthralgia disease activity is assessed by a disease-specific daily health assessment form (FXII-associated Cold autoinflammatory Syndrome daily Health assessment form; FACAS-DHAF; scale 0=no symptoms to 10=max. of symptoms)
Change in headache disease activity score as assessed by daily health assessment form (DHAF) questionnaire following lanadelumab treatment | weeks 9 to 12 and weeks 24 to 28, each compared to weeks -4 to -1 (baseline)
  Patient-reported headache disease activity is assessed by a disease-specific daily health assessment form (FXII-associated Cold autoinflammatory Syndrome daily Health assessment form; FACAS-DHAF; scale 0=no symptoms to 10=max. of symptoms)
Change in total disease activity score as assessed by daily health assessment form (DHAF) questionnaire following lanadelumab Treatment over Long-term use | weeks 24 to 28 compared to weeks -4 to -1 (baseline)
  Patient-reported total disease activity is assessed by a disease-specific daily health assessment form (FXII-associated Cold autoinflammatory Syndrome daily Health assessment form; FACAS-DHAF; scale 0=no symptoms to 50=max. of symptoms
Change in inflammation markers following lanadelumab Treatment | from Baseline to week 12 and week 28
  Assessment of CRP levels
Change in inflammation markers following lanadelumab Treatment | from Baseline to week 12 and week 28
  Assessment of ESR levels
Change in inflammation markers following lanadelumab Treatment | from Baseline to week 12 and week 28
  Assessment of SAA levels
Change in inflammation markers following lanadelumab Treatment | from Baseline to week 12 and week 28
  Assessment of S100 A8/9 levels
Change in dermatology-specific quality-of-life following lanadelumab Treatment | from Baseline to week 12 and week 28
  assessed by Dermatology Life Quality Index (DLQI); scale 0=no impairment to 30=max. impairment
Changes in generic Health-related quality-of-life | from Baseline to week 12 and week 28
  assessed by 36-Item Short Form Health Survey (SF-36); scale 0=max. impairment to 100=no impairment (best Quality of life)
Incidence of of Treatment-emergent adverse Events, abnormal physical examination, abnormal Routine safety laboratory assessments, abnormal vital signs (safety and tolerability) | from Baseline to end of study (week 36 follow-up)
  Safety of lanadelumab Treatment is assessed by physical examination, routine safety laboratory assessments, vital signs, and adverse Event reporting.
Change in physician global assessment following lanadelumab Treatment as assessed by verbal rating scale | from Baseline to week 12 and week 28
  Verbal Rating scale assesses overall Symptoms from 0-10 (0=no symptoms; 10=very severe symptoms)
Changes of plasma levels of potential biomarkers following Lanadelumab treatment | from Baseline to week 28
  Potential biomarkers include Plasma FXII Levels
Changes of plasma levels of potential biomarkers following Lanadelumab treatment | from Baseline to week 28
  Potential biomarkers include Plasma prekallikrein Levels
Changes of plasma levels of potential biomarkers following Lanadelumab treatment | from Baseline to week 28
  Potential biomarkers include Plasma cHMWK Levels
Changes of plasma levels of potential biomarkers following Lanadelumab treatment | from Baseline to week 28
  Potential biomarkers include IL-1ß release from donor PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Krause, Prof., Principal Investigator — Charité University, Berlin, Germany
Locations (1):
- Charite University, Berlin, Germany, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No